CLINICAL TRIAL: NCT04632654
Title: A Motion Exergaming Approach to Promote Self-Managing Fatigue and Pain After Head and Neck Cancer Treatment
Brief Title: A Motion Exergaming Approach for Symptom Management: HNC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hsiao-Lan Wang, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY000062; 1R01CA244947-01 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-11-17 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAfitME (Experimental): For 6 weeks, the experimental (PAfitME) group will receive the PAfitME intervention.
  Interventions: Behavioral: A personalized Physical Activity intervention with fitness graded Motion Exergames (PAfitME)
- Attention Control (No Intervention): For 6 weeks, the attention control group will receive National Cancer Institute-based survivorship education and exergame equipment (Nintendo Switch).

INTERVENTIONS:
Behavioral: A personalized Physical Activity intervention with fitness graded Motion Exergames (PAfitME) — A total of 7 weekly intervention sessions will occur in a period of 6 weeks. Week 0 is a setup session conducted at the participant's home, including equipment set up, safety instruction, personalized exergame prescription development, exergame physical activity practice, discussion of barriers and strategies, and Q&A session. Weeks 1 and 2 are coaching sessions delivered by the interventionist using the FaceTime application in iPad, including exergame minutes and prescription review, exergame physical activity practice, discussion of barriers and strategies, and Q&A session. Week 3 is a progress session conducted at the participant's home. The personalized exergame prescription will be adjusted. This session also will include exergame minutes review, exergame physical activity practice, discussion of barriers and strategies, and Q&A session. Weeks 4 and 5 are the same as weeks 1 and 2. Week 6 is the final session. Exergame platform will be picked up at the participant's home.
  Arms: PAfitME

SUMMARY:
This overall objective of the RCT is to test an intervention to overcome the PA barriers for head and neck cancer (HNC) patients during the first 6 months after their treatment. PAfitME stands for a personalized Physical Activity intervention with fitness graded Motion Exergames. PAfitME is delivered via a tested mix of FaceTime calls and home visits, uses commercially available exergaming platforms (Nintendo Switch). We propose the following specific aims: (1) When compared to an attention control group, determine the effect of PAfitME on fatigue and musculoskeletal pain at week 6, when controlling for age and sex; (2) when compared to an attention control group, determine the effect of PAfitME on functional status and QOL at week 6, when controlling for age and sex; and (3) explore if PA self-efficacy, PA enjoyment, and exergame minutes mediate the effect of PAfitME on fatigue and musculoskeletal pain. This study will evaluate 150 post-treatment (radiation, chemotherapy, or chemoradiation) HNC patients in an RCT with an attention control. For 6 weeks, the experimental (PAfitME) group will receive the PAfitME intervention, and the attention control group will receive NCI-based survivorship education and exergame equipment. For Aims 1 and 2, using an intention-to-treat framework, we will fit a series of linear mixed effects models with each of the outcome variables. For Aim 3, we will conduct our exploratory analyses in ml_mediation (STATA 15), which will compute direct and indirect effects for multi-level data.

DETAILED DESCRIPTION:
Among head and neck cancer (HNC) patients, 92% report fatigue and 73% have pain. A 10% increase in fatigue or pain is associated with a 10-25% reduction in HNC survival. During the critical transition period from the end of active treatment to 6 months post-treatment, untreated physical symptoms negatively impact functional status (ADL) and quality of life (QOL). Fatigue and musculoskeletal pain are known to improve in response to physical activity (PA). However, 51% of HNC survivors rarely engage in any type of PA because of complicated PA barriers. Our overall objective is to test an intervention to overcome these PA barriers for HNC patients during the critical transition period to self-management. PAfitME, a personalized Physical Activity intervention with fitness graded Motion Exergames, is a telehealth program built on Social Cognitive Theory and the exercise principle of adaptation. PAfitME, delivered via a tested mix of FaceTime calls and home visits, uses commercially available exergaming platforms (Wii Fit and Xbox Kinect). We propose the following specific aims: (1) When compared to an attention control group, determine the effect of PAfitME on fatigue and musculoskeletal pain at week 6, when controlling for age and sex; (2) when compared to an attention control group, determine the effect of PAfitME on functional status and QOL at week 6, when controlling for age and sex; and (3) explore if PA self-efficacy, PA enjoyment, and exergame minutes mediate the effect of PAfitME on fatigue and musculoskeletal pain. This study will evaluate 150 post-treatment (radiation, chemotherapy, or chemoradiation) HNC patients in an RCT with an attention control. For 6 weeks, the experimental (PAfitME) group will receive the PAfitME intervention, and the attention control group will receive NCI-based survivorship education and exergame equipment. For Aims 1 and 2, using an intention-to-treat framework, we will fit a series of linear mixed-effects models with each of the outcome variables. For Aim 3, we will conduct our exploratory analyses in ml_mediation (STATA 15), which will compute direct and indirect effects for multi-level data. This study aligns with the NCI Cancer Moonshot goal to minimize cancer treatment-associated side effects and the key recommendation in the National Comprehensive Cancer Network Clinical Guidelines of the need for evidence-based non- pharmacological fatigue/pain treatments (National Priority).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, patients must be:

1. diagnosed with head and neck cancer (Tumor sites in the head and neck area);
2. 18 years or older;
3. able to understand English;
4. able to communicate;
5. have a Karnofsky Performance Status (KPS) score of >= 60%;
6. be cleared by their provider to resume low to moderate intensity PA;
7. have fatigue or pain of ≥moderate severity; and

A KPS score of >= 60% has been used in previous exercise trials in the HNC population. This is equal to ECog scores ≤ 2.

Moderate fatigue or pain severity is defined as a worst score in the past week of >= 4 on a 0-10 scale.

Patients receiving immunotherapy are not excluded from participating in the study.

Exclusion Criteria:

Patients will be excluded if they

1. are hospitalized;
2. are in hospice care;
3. have a history of seizures or loss of consciousness; or
4. are cognitively impaired, defined as making ≥3 errors on a validated 6-item cognitive screener (3 items identifying the current year, month, and day; 3 items recalling 3 pre-selected objects).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0-Fatigue (NIH Common Data Elements [CDE]). | Baseline and Week 6
  In the PROMIS Short Form v1.0-Fatigue, the 6 items ask about fatigue status, including fatigue severity and fatigue distress in the past 7 days. The scale ranges from 1 to 5. The higher the score, the worse the symptom. The mean score of 6 items will be calculated in the analysis to test the changes from baseline to week 6.
Musculoskeletal Pain will be measured by the PROMIS Short Form v.1.0-Pain Intensity (CDE). | Baseline and Week 6
  In the PROMIS Short Form v1.0-Pain, the 3 items ask about pain intensity in the past 7 days. The scale ranges from 1 to 5. The higher the score, the worse the symptom. The mean score of 3 items will be calculated in the analysis to test the changes from baseline to week 6.

SECONDARY OUTCOMES:
Subjective Functional Status will be measured by the self-report Lawton Instrumental Activities of Daily Living Scale (IADL). | Baseline and Week 6
  In the IADL, the 8-item IADL measures dependence/independence of 8 daily activities. Participants will respond based on their highest level of independence for that activity. The total score ranges from 8 to 31. The higher the score, the better the function. The toal score of 8 items will be calculated in the analysis to test the changes from baseline to week 6.
Objective Functional Status will be measured by 2-minute walk test. | Baseline and Week 6
  The 2-minute walk measures distance (in meters) walked in 2 minutes. The distance in meters will will be calculated in the analysis to test the changes from baseline to week 6.
Objective Functional Status will be measured by combined grip sum. | Week 0 and Week 6
  Combined grip sum is calculated by "[left hand grip strength maximum + right hand grip strength maximum] ÷ body weight". It levels out the dominant hand effect (by using the sum of left hand and right hand strength) and represents the ratio of hand muscle strength and body weight. Hand grip strength will be measured by Jamar hydraulic hand dynamometer (Jamar Technologies, Inc., Hatfield, PA).The combined grip sum will be calculated in the analysis to test the changes from baseline to week 6.
Objective Functional Status will be measured by upper extremity range of motion (ROM). | Week 0 and Week 6
  Upper extremity ROM is upper extremity flexibility and includes shoulder abduction, shoulder forward flexion, neck forward flexion, neck extension, neck lateral flexion, and neck lateral rotation. The ROM will be measured by a plastic 12" goniometer 360 degree (Szy Holdings LLC, Brooklyn, NY). The degrees of range of motion will be calculated in the analysis to test the changes from baseline to week 6.
Objective Functional Status will be measured by chair sit and reach. | Week 0 and Week 6
  Chair sit and reach is to measure lower extremity flexibility. The participant sits on a chair with one foot flat on the floor to support the balance and the other leg extended forward with knee straight, heel on the floor, and ankle bent at 90º. With one hand on top of the other, the participant reaches forward toward the toes by bending at the hip. The distance between the tip of the fingertips and the toes is measured. If the fingertips touch the toes, the score is zero. If they do not touch, the distance between the fingers and the toes (a negative score) is measured; if they overlap, the overlap distance is measured (a positive score). The distance in positive or negative centImeters (cm) will be calculated in the analysis to test the changes from baseline to week 6.
Objective Functional Status will be measured by Timed up and go. | Week 0 and Week 6
  Timed up and go requires participants to stand up from a chair, walk 3 meters, turn around, walk back to the chair and sit down. The result of the test is the time from standing up from the chair to sitting back on the same chair. The time in seconds will be calculated in the analysis to test the changes from baseline to week 6.
Quality of Life will be measured using the Functional Assessment of Chronic Illness Therapy-Head and Neck Scale, version 4 (FACIT-H&N). | Week 0 and Week 6
  FACIT-H&N includes a 28-item general scale and a 12-item HNC scale. The scale ranges from 0 to 4. The greater the score, the better the quality of life. The mean scores of the 28-item general scale and 12-item HNC scale will be calculated in the analysis to test the changes from baseline to week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Lan Wang, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No